CLINICAL TRIAL: NCT03068481
Title: A Phase I Clinical Study of KDT-3594 in Healthy Adult Males and Patients With Parkinson's Disease
Brief Title: Clinical Study of KDT-3594 in Healthy Adult Males and Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KDT1102
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Healthy volunteer part -Multiple dose: Parallel, Healthy volunteer part -Single dose and Patient part: Single Group
Who Masked: Participant
Masking Description: Healthy volunteer part -Multiple dose: Participant, Healthy volunteer part -Single dose and Patient part: No Masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy volunteer part -Single dose (Experimental): Single oral dose of KDT-3594
  Interventions: Drug: KDT-3594
- Healthy volunteer part -Multiple dose (Experimental): Multiple oral doses of KDT-3594
  Interventions: Drug: KDT-3594
- Healthy volunteer part -Placebo (Placebo Comparator): Multiple oral doses of Placebo
  Interventions: Drug: Placebo
- Patient part -Single dose (Experimental): Single oral dose of KDT-3594
  Interventions: Drug: KDT-3594
- Patient part -Multiple dose (Experimental): Multiple oral doses of KDT-3594
  Interventions: Drug: KDT-3594

INTERVENTIONS:
Drug: KDT-3594 — Oral administration
  Arms: Healthy volunteer part -Multiple dose; Healthy volunteer part -Single dose; Patient part -Multiple dose; Patient part -Single dose
Drug: Placebo — Oral administration
  Arms: Healthy volunteer part -Placebo

SUMMARY:
The purpose of this study in healthy adult males is to investigate safety and pharmacokinetics of single and multiple oral doses of KDT-3594.

The purpose of this study in patients with Parkinson's disease is to investigate safety and pharmacokinetics of single and multiple oral doses of KDT-3594. The exploratory efficacy of KDT-3594 will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer part

  * Healthy Japanese males aged 20 to 35 years, inclusive
* Patient part

  * Patients who are diagnosed with Parkinson's disease according to UK Parkinson's Disease society brain bank clinical diagnostic criteria
  * Patients with Parkinson's disease in Stages 1 to 3 on the Modified Hoehn and Yahr Scale
  * Male patients with Parkinson's disease aged 20 to 74 years inclusive, post-menopausal female patients with Parkinson's disease aged 50 to 74 years inclusive

Exclusion Criteria:

* Healthy volunteer part

  * Subjects with any abnormal findings in physical examination vital signs, 12-lead ECG, clinical laboratory tests, ophthalmic examinations and electroencephalography
* Patient part

  * Patients who are suspected any parkinsonism except for idiopathic Parkinson's disease
* Healthy volunteer part and patient part

  * Subjects who do not agree to avoid dangerous works such as driving, mechanical operation and high-place work until completion of the follow-up examination

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | Up to 15 days after last administration
Plasma pharmacokinetic parameter of KDT-3594 and main metabolites: Cmax | Up to 336 hours after last administration
Plasma pharmacokinetic parameter of KDT-3594 and main metabolites: AUC | Up to 336 hours after last administration

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) score (Only patient part) | Up to 336 hours after last administration

CONTACTS AND LOCATIONS:
Locations (1):
- Kyushu and Other Regions, Japan